CLINICAL TRIAL: NCT06103981
Title: Acute Liver Injury in Patients With Pneumonia and Its Impact on Hospital Stay and Outcome
Brief Title: Acute Liver Injury in Patients With Pneumonia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Beshoy Yousef Boles Abdelmalak, Resident, Assiut University
Other Study IDs: Acute Liver Injury
Record Dates: First submitted 2023-08-12; First posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Acute Liver Injury; Pneumonia
Keywords: Acute Liver Injury; pneumonia; Covid19
MeSH Terms: conditions — Pneumonia; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: About 88 patients having pneumonia and developed acute liver injury That need observation of the outcome and hospital stay to evaluate acute liver injury impact
  Interventions: Other: Acute Liver Injury
- Group B: About 88 patients having pneumonia but did not develop acute liver injury that need observation of the outcome and hospital stay
  Interventions: Other: Acute Liver Injury

INTERVENTIONS:
Other: Acute Liver Injury — To evaluate the impact of acute liver injury in patients with pneumonia on hospital stay and outcome.

SUMMARY:
Acute liver injury (ALI) is defined as an acute derangement in liver function tests associated with liver-related coagulopathy, in the absence of underlying chronic liver disease.

A subset progress to acute liver failure ,Acute liver failure represent a more severe liver injury results in hepatic encephalopathy

DETAILED DESCRIPTION:
Acute liver injury is associated with a spectrum of haemostatic changes, including thrombocytopenia and reduced platelet function, reduced plasma levels of many coagulation factors such as factor (F)VII and increased levels of FVIII .

Pneumonia is an acute inflammation of the lower respiratory tract. Lower respiratory tract infection is a major cause of mortality worldwide .Pneumonia is most common at the extremes of life.

In adults, pneumonia can be broadly classified, on the basis of chest radiographic appearance, into lobar pneumonia, bronchopneumonia and pneumonia producing an interstitial pattern.

There is lack of data regarding outcome and hospital stay in patients with pneumonia who develop acute liver injury.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pneumonia that developed Acute Liver Injury
2. Covid 19 pneumonia
3. Patients With acute liver injury only.

Exclusion Criteria:

1. Cancer
2. Immunocompromised patients i.e HIV patients and patients who take immunosuppressive medications.
3. Patients who younger than 18 yrs old
4. pregnancy

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with pneumonia in hospital ward or critical care
Sampling Method: Non-Probability Sample
Enrollment: 176 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2025-01-10 (Estimated); Study Completion 2025-03-10 (Estimated)

PRIMARY OUTCOMES:
Impact of Acute liver injury due to Pneumonia | From Hospital admission date to Two Months
  Analysis the impact of acute liver injury related to patients with pneumonia on hospital stay (measured by days spent in the hospital).

SECONDARY OUTCOMES:
Patients with Pneumonia only | From Hospital admission date to Two Months
  To evaluate the Patients with Pneumonia either developed acute liver injury or not, On Hospital Stay

CONTACTS AND LOCATIONS:
Overall Officials: Zain Elabdeen Ahmed, Professor, Study Chair — Assuit Faculty of Medicine
Locations (1):
- Faculty Of Medicine, Asyut, Egypt